CLINICAL TRIAL: NCT01391130
Title: Randomized, Multicenter, Open-label, Active-Controlled, Phase 2 Study of LY2510924 and Sunitinib Versus Sunitinib in Patients With Metastatic Renal Cell Carcinoma
Brief Title: A Study of LY2510924 and Sunitinib in Patients With Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Terminated due to Insufficient Efficacy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14241; I2V-MC-CXAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-06

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma
Keywords: Cancer; Tumor; Metastasis
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Neoplasms; Neoplasm Metastasis | interventions — LY2510924; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2510924 + Sunitinib (Experimental): LY2510924: 20 milligram administered subcutaneously once daily, given every day of the 6 week cycle. Sunitinib: 50 milligram administered orally once daily, on a schedule of 4 weeks on treatment followed by 2 weeks off treatment. Treatment cycles will continue until disease progression, unacceptable toxicity, or another withdrawal criterion is met.
  Interventions: Drug: LY2510924; Drug: Sunitinib
- Sunitinib (Active Comparator): 50 milligram administered orally once daily, on a schedule of 4 weeks on treatment followed by 2 weeks off treatment. Treatment cycles will continue until disease progression, unacceptable toxicity, or another withdrawal criterion is met.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: LY2510924 — Administered subcutaneously
  Arms: LY2510924 + Sunitinib
Drug: Sunitinib — Administered orally

SUMMARY:
To compare the progression free survival of LY2510924 plus sunitinib therapy versus sunitinib in the first-line setting for patients with metastatic clear-cell renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of histologically confirmed renal cell carcinoma (RCC) with metastases with a component of clear (conventional) cell histology
* A diagnosis of metastatic renal cell carcinoma (RCC) and have not received prior treatment with systemic (adjuvant or neoadjuvant) therapy for renal cell carcinoma (RCC) (including targeted therapy such as tyrosine kinase inhibitors or bevacizumab, immunotherapy, chemotherapy, hormonal, or investigational therapy)
* Evidence of measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Computed tomography (CT) or magnetic resonance imaging (MRI) should be performed within 4 weeks prior to study entry
* Participants who have or have not had their primary tumor removed by nephrectomy are allowed. Participants who have not had a nephrectomy should not be considered to need a nephrectomy as part of their overall therapy at the time of enrollment
* Performance status score of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Adequate bone marrow, liver, and renal function, as assessed by the following laboratory requirements, to be conducted within seven days prior to treatment: (upper limit of normal/lower limit of normal [ULN/LLN])

  * hemoglobin (greater than) >8.0 g/dL (grams per deciliter)
  * absolute neutrophil count (ANC) (greater than or equal to) ≥1.5 × 10^9/L (liter)
  * platelet count (greater than or equal to) ≥100 × 10^9/L (liter)
  * total bilirubin (less than or equal to) ≤ 1.5 × ULN (upper limit of normal)
  * serum creatinine (less than or equal to) ≤2 × ULN (upper limit of normal)
  * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) (less than or equal to) ≤2.5 × ULN (upper limits of normal) [or (less than or equal to) ≤5 × ULN (upper limits of normal) for patients with liver involvement of their cancer]
  * Prothrombin Time (PT) or International Normalized Ratio (INR) and activated Partial Thromboplastin Time (aPTT) (less than or equal to) ≤1.5 x ULN (upper limit of normal)
* For women: Must be surgically sterile (surgical procedure: bilateral tubal ligation, hysterectomy, bilateral oophorectomy), post-menopausal (at least 12 consecutive months of amenorrhea), or have a negative pregnancy test. Women of childbearing potential should be compliant with a medically approved contraceptive regimen (intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after the treatment period; must have a negative serum pregnancy test within 7 days before study enrollment, and must not be breastfeeding
* For men: Must be surgically sterile or compliant with a contraceptive regimen during and for 3 months after the treatment period
* Estimated life expectancy of at least 12 weeks
* Provide written informed consent/assent prior to any study-specific procedures
* No prior malignancies with the exception of stage 1 cancers definitively treated, carcinoma in situ (any primary site), treated non-melanoma skin cancer, superficial bladder tumors (Ta, Tis, and T1) or any cancer curatively treated 5 or more years prior to study entry
* Capable and willing to learn to self-administer LY2510924, or have a caregiver who is willing to learn and able to administer LY2510924 by subcutaneous (SC) injection and are able to swallow tablets
* Left ventricular ejection fraction (LVEF) greater than or equal to LLN as defined by the institution performing the scan, as assessed by Multiple Gated Acquisition (MUGA) scan, or from echocardiogram to be performed within 28 days prior to start of treatment

Exclusion Criteria:

* Received prior treatment with sunitinib or LY2510924
* Received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* History of active cardiovascular disease within the previous 12 months, including any of the following:

  * Myocardial infarction
  * Unstable angina
  * Coronary artery/peripheral artery bypass graft
  * Congestive heart failure
  * Malignant hypertension
  * Cerebrovascular accident or transient ischemic attack
  * Symptomatic cardiac arrhythmias (Patients with chronic, stable, rate- controlled atrial fibrillation are eligible)
* Exhibit uncontrolled hypertension ( [greater than] >150/100 [millimeters of mercury] mm/Hg despite optimal medical therapy), or history of poor compliance with antihypertensive treatment
* Evidence of bleeding diathesis, National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 hemorrhage (less than) <4 weeks of starting the study treatment, coagulopathy, or thromboembolic event
* Significant surgery (less than) <4 weeks of starting study treatment or a minor surgical procedure (less than) < 7 days prior to study treatment (Placement of a portacath or other venous access device does not require a waiting period)
* Suffer from medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to any agent given in association with this trial
* Prior palliative radiotherapy to metastatic lesion(s) is/are permitted, provided there is at least 1 measurable lesion that has not been irradiated. Radiotherapy must have been completed (greater than) >2 weeks prior to starting study treatment, and radiation-related side effects must have resolved
* Pregnant or lactating women
* Impairment of the gastrointestinal (GI) function or GI disease that may significantly alter the absorption of sunitinib
* Current or recent (within 10 days of first dose of study treatment) daily use of aspirin ( [greater than] >325 [milligram] mg/day )
* Serious nonhealing wounds, acute or nonhealing ulcers, or bone fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- United States (21):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norwich, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newark, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pensacola, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lawrenceville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bridgeton, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morristown, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lawton, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Worth, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

REFERENCES:
- [Derived] Hainsworth JD, Reeves JA, Mace JR, Crane EJ, Hamid O, Stille JR, Flynt A, Roberson S, Polzer J, Arrowsmith ER. A Randomized, Open-Label Phase 2 Study of the CXCR4 Inhibitor LY2510924 in Combination with Sunitinib Versus Sunitinib Alone in Patients with Metastatic Renal Cell Carcinoma (RCC). Target Oncol. 2016 Oct;11(5):643-653. doi: 10.1007/s11523-016-0434-9. PMID 27154357

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who died (any cause) or had disease progression at the time the primary analysis were considered to be study completers.
Period: Overall Study
Arm/Group | LY2510924 + Sunitinib | Sunitinib
Started | 73 | 37
Received At Least One Dose of Study Drug | 72 | 36
Completed | 67 | 31
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Physician Decision | 2 | 3
Not completed — Did not Receive Drug | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2510924 + Sunitinib | Sunitinib | Total
Number analyzed (Participants) | 72 | 36 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.51 (11.332) | 64.21 (9.474) | 64.41 (10.705)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 12 | 36
  Male | 48 | 24 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 71 | 34 | 105
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 68 | 34 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72 | 36 | 108

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from date of study Randomization to the first date of objectively determined progressive disease(PD) or death from any cause defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.0).PD was defined as at least a 20% increase in the sum of the diameters of target lesions,taking as reference the smallest sum on study(including the baseline sum if that is the smallest).In addition to the relative increase of 20%,the sum must also demonstrate an absolute increase of at least 5 mm.The appearance of one or more new lesions was also considered PD.For participants still alive at the time of analysis and without evidence of tumor progression,PFS would be censored at the date of the most recent objective progression-free observation.For participants who receive subsequent anticancer therapy prior to objective disease progression or death,PFS was censored at the date of the last objective progression-free observation prior to the date of subsequent therapy.
Time Frame: Randomization to Measured Progressive Disease or Date of Death From Any Cause (Up to 67 Months)
Population: All participants who received at least one dose of study drug. Participants censored were LY2510924 + Sunitinib = 16 and Sunitinib=12.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LY2510924 + Sunitinib | Sunitinib
Number analyzed (Participants) | 72 | 36
Months | 8.08 [5.52 to 10.64] | 12.25 [2.66 to 20.01]
Statistical Analysis 1: Comparison: LY2510924 + Sunitinib vs Sunitinib; Test type: Superiority; p = 0.4318, Log Rank; Hazard Ratio (HR) = 1.2149, 95% CI 2-sided [0.7462 to 1.9779]

2. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) (Overall Response Rate[ORR])
Description: ORR is defined as the number of participants with a best response of CR and PR defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) criteria. CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Tumor marker results must have normalized. PR is defined as at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.The appearance of one or more new lesions is also considered progression.
Time Frame: Baseline to Date of Tumor Response or Measured Progressive Disease or Date of Death from any Cause ((Up to 67 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LY2510924 + Sunitinib | Sunitinib
Number analyzed (Participants) | 72 | 36
percentage of participants | 31.9 [21.17 to 42.71] | 38.9 [22.96 to 54.81]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of study randomization to the date of death from any cause. For participants who were still alive as of the data cut-off date, OS time will be censored on the date of the participant's last contact (last contact for participants in post-discontinuation = last known alive date in mortality status).
Time Frame: Randomization to Date of Death from Any Cause (Up to 67 Months)
Population: All participants who received at least one dose of study drug. Participants censored were LY2510924 + Sunitinib=19 and Sunitinib=10.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LY2510924 + Sunitinib | Sunitinib
Number analyzed (Participants) | 72 | 36
months | 24.18 [13.90 to 35.19] | 23.82 [11.60 to 43.86]

4. Secondary Outcome: Duration of Overall Response (DOR)
Description: DOR was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause. Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) criteria. CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Tumor marker results must have normalized. PR is defined as at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD)is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Date of First Response to Date of Progressive Disease (Up to 67 Months)
Population: All participants who received at least one dose of study drug. Participants censored were LY2510924 + Sunitinib=7 and Sunitinib=7.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LY2510924 + Sunitinib | Sunitinib
Number analyzed (Participants) | 72 | 36
Months | 11.30 [5.36 to 16.99] | 12.42 [3.15 to NA] — The data were not evaluable for the upper confidence interval.

5. Secondary Outcome: Duration of Complete Response
Description: Duration of complete response is defined as the time from the date when the measurement criteria are met for complete response until the date of first observation of objective disease progression (taking as reference for PD the smallest measurements recorded since the treatment started). CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Tumor marker results must have normalized. Progressive Disease (PD)is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Date of Complete Response to the Date of Progressive Disease (Up to 67 Months)
Population: All participants who received at least one dose of study drug who had CR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LY2510924 + Sunitinib | Sunitinib
Number analyzed (Participants) | 0 | 1
months |  | 10 [NA to NA] — Only one participant had CR.

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug.
Arm/Group | LY2510924 + Sunitinib | Sunitinib
Serious Adverse Events (participants affected / at risk) | 31/72 | 10/36
Other Adverse Events (participants affected / at risk) | 70/72 | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2510924 + Sunitinib (N=72) | Sunitinib (N=36)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Pancreas infection (Infections and infestations) | 1 (1) | 0 (0)
Peridiverticular abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (2)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Spinal operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2510924 + Sunitinib (N=72) | Sunitinib (N=36)
Anaemia (Blood and lymphatic system disorders) | 26 (95) | 7 (10)
Leukocytosis (Blood and lymphatic system disorders) | 5 (6) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (4) | 5 (8)
Neutropenia (Blood and lymphatic system disorders) | 6 (22) | 4 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 20 (57) | 9 (12)
Hypothyroidism (Endocrine disorders) | 11 (11) | 3 (3)
Vision blurred (Eye disorders) | 5 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (9) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 1 (1)
Constipation (Gastrointestinal disorders) | 16 (19) | 6 (10)
Diarrhoea (Gastrointestinal disorders) | 28 (55) | 18 (39)
Dry mouth (Gastrointestinal disorders) | 6 (7) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 4 (6)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (3)
Flatulence (Gastrointestinal disorders) | 4 (5) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (8) | 2 (4)
Glossodynia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 5 (9) | 1 (1)
Nausea (Gastrointestinal disorders) | 35 (50) | 18 (33)
Oral pain (Gastrointestinal disorders) | 6 (6) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 15 (19) | 7 (11)
Vomiting (Gastrointestinal disorders) | 18 (32) | 8 (14)
Asthenia (General disorders) | 9 (10) | 0 (0)
Chest pain (General disorders) | 5 (5) | 1 (1)
Chills (General disorders) | 6 (7) | 0 (0)
Fatigue (General disorders) | 50 (96) | 20 (37)
Injection site pruritus (General disorders) | 6 (6) | 0 (0)
Injection site reaction (General disorders) | 6 (6) | 0 (0)
Mucosal inflammation (General disorders) | 17 (25) | 10 (15)
Oedema (General disorders) | 3 (3) | 2 (2)
Oedema peripheral (General disorders) | 17 (27) | 6 (8)
Pain (General disorders) | 3 (3) | 2 (13)
Pyrexia (General disorders) | 10 (10) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 9 (11) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 2 (2)
Urinary tract infection (Infections and infestations) | 8 (16) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 6 (7) | 2 (3)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 7 (8) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 5 (5) | 2 (2)
Blood creatinine increased (Investigations) | 5 (6) | 5 (7)
Weight decreased (Investigations) | 12 (15) | 9 (13)
Weight increased (Investigations) | 2 (4) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 17 (26) | 8 (14)
Dehydration (Metabolism and nutrition disorders) | 12 (19) | 5 (12)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (4) | 3 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (8) | 1 (1)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (23) | 2 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (9) | 4 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 17 (20) | 7 (11)
Dysgeusia (Nervous system disorders) | 23 (27) | 11 (14)
Headache (Nervous system disorders) | 10 (14) | 6 (6)
Anxiety (Psychiatric disorders) | 9 (11) | 3 (4)
Confusional state (Psychiatric disorders) | 4 (6) | 1 (3)
Depression (Psychiatric disorders) | 7 (7) | 2 (2)
Insomnia (Psychiatric disorders) | 7 (9) | 5 (7)
Dysuria (Renal and urinary disorders) | 4 (4) | 1 (1)
Haematuria (Renal and urinary disorders) | 8 (9) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0/24 (0) | 1/12 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (19) | 7 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (9) | 3 (4)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 12 (38) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (5)
Rash (Skin and subcutaneous tissue disorders) | 19 (28) | 4 (6)
Skin lesion (Skin and subcutaneous tissue disorders) | 5 (7) | 1 (1)
Hypertension (Vascular disorders) | 17 (26) | 12 (18)

LIMITATIONS AND CAVEATS:
Study Terminated due to Insufficient Efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days